CLINICAL TRIAL: NCT03592888
Title: Pilot Study of Mature Dendritic Cell Vaccination Against Mutated KRAS in Patients With Resectable Pancreatic Cancer
Brief Title: DC Vaccine in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04218
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma; Cancer vaccine; Dendritic cell vaccine; Mutant KRAS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Experimental): All subjects will receive the vaccine and be followed per the schedule of procedures.
  Interventions: Drug: mDC3/8-KRAS Vaccine

INTERVENTIONS:
Drug: mDC3/8-KRAS Vaccine — Mature dendritic cell (mDC3/8) vaccine (primer and booster) in subjects with resected pancreatic adenocarcinoma

SUMMARY:
This research study is designed to evaluate the effects of a dendritic cell (kind of white blood cell) vaccine for pancreatic cancer.

DETAILED DESCRIPTION:
This is a single arm open label trial that will assess the safety and tolerability of mature dendritic cell (mDC3/8) vaccine (primer and booster) in subjects with resected pancreatic adenocarcinoma.

Eligible patients that provide written informed consent will undergo apheresis to collect blood mononuclear cells for vaccine production approximately 1 week prior to vaccine infusion. Each study subject will receive cyclophosphamide 300mg/m^2 intravenously 3 to 4 days prior to the vaccine dose to deplete regulatory T cells. For each vaccine dose, all subjects will receive autologous dendritic cells pulsed with mutant KRAS peptides corresponding to the subject's specific tumor mutation and human leukocyte antigen type. On Day 1, the subject will receive the primer vaccine dose; this will be followed by one booster vaccine dose approximately 8 weeks later. Peripheral blood will be taken weekly, and a second apheresis procedure will be performed at the end of study to monitor the immune response to the vaccine. Information will be gathered from usual clinic visits for approximately 1 year following the End of Treatment Study Visit to evaluate for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed KRAS(G12D-), KRAS(G12V-), KRAS(G12R-) or KRAS(G12C-mutated) pancreatic ductal adenocarcinoma who are at high risk of relapse and have no evidence of disease.
* Expression of one or more of the following HLA class I alleles: HLA-A02, HLA-A03, HLA-A11, HLA-B07 and HLA-C08.
* Male or female, age 18+
* ECOG performance status 0-1
* Certain required laboratory values, performed within 14 days prior to consent
* Subjects of reproductive potential must agree to use a medically accepted birth control method during the trial and for at least two months following the trial.
* Provide written informed consent

Exclusion Criteria:

* Prior treatment with more than two lines of cytotoxic chemotherapy. Radiotherapy is not considered a line of therapy.
* Prior malignancy (except non-melanoma skin cancer) within 3 years.
* Pregnant or nursing women.
* Concurrent treatment with systemic immunosuppressants, including corticosteroids (e.g prednisone), calcineurin inhibitors (e.g tacrolimus, cyclosporine), antiproliferative agents (e.g mycophenolate mofetil, azathioprine) within 2 weeks of eligibility confirmation. Local (inhaled or topical) steroids or replacement dose prednisone (≤ 10 mg daily) are permitted.
* Known chronic viral infections including hepatitis B, hepatitis C, and HIV.
* Known allergy to eggs.
* Prior history of uveitis or autoimmune inflammatory eye disease.
* Uncontrolled intercurrent illness.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Safety and side effects of vaccine per CTCAE 4.0 | At time of consent through 30 days after the subject's last DC vaccine

SECONDARY OUTCOMES:
Immune response measuring increased numbers of peptide specific T cells as calculated by the peptide-MHC multimer assay. | Day 1 through week 12
Disease Free Survival | 30 days following second vaccine through study completion approximately 12 months after the first DC vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Mark O'Hara, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bear AS, Nadler RB, O'Hara MH, Stanton KL, Xu C, Saporito RJ, Rech AJ, Baroja ML, Blanchard T, Elliott MH, Ford MJ, Jones R, Patel S, Brennan A, O'Neil Z, Powell DJ Jr, Vonderheide RH, Linette GP, Carreno BM. Natural TCRs targeting KRASG12V display fine specificity and sensitivity to human solid tumors. J Clin Invest. 2024 Sep 17;134(21):e175790. doi: 10.1172/JCI175790. PMID 39287991